CLINICAL TRIAL: NCT04947072
Title: Comparison Between Erector Spinae Plane Block and Spinal as Surgical Anesthesia and Analgesia in Percutaneous Nephrolithotomy Patient : Conversion to General Anesthesia, Interleukin-6, Postoperative Pain and Opioid Consumption
Brief Title: Erector Spinae Plane Block and Spinal Anesthesia for Supine Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Pryambodho Pryambodho, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes106
Record Dates: First submitted 2021-06-26; First posted 2021-07-01 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Incidence Conversion to General Anesthesia, Interleukin-6, Total Tramadol Consumption and Pain Score After Surgery
Keywords: Erector Spinae Plane Block; Percutaneous Nephrolithotomy; Interleukin-6, Effectiveness; Tramadol patient controlled analgesia; Visual analog scale
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): Patient will receive single-shot ultrasound-guided erector spinae plane block at the level of T9 on the side which will be operated on.
  Interventions: Procedure: Erector Spinae Plane Block; Procedure: Spinal anesthesia
- Spinal Anesthesia (Active Comparator): Patient will receive spinal anesthesia at the level of L3-L4 or L4-L5
  Interventions: Procedure: Erector Spinae Plane Block; Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — The block will be performed at the level of T9 on the site that will be operated and patient will be given Bupivacaine isobaric 0.5% 25 ml with epinephrine 1:200.000
Procedure: Spinal anesthesia — Patient will be given bupivacaine hyperbaric 0.5% 16-18 mg at the level of L3-L4 or L4-L5

SUMMARY:
This study aimed to compare the Effectiveness of Erector Spinae plane block to Spinal as a surgical anesthesia and analgesia in Percutaneous Nephrolithotomy patient

DETAILED DESCRIPTION:
Thirty subjects (who meet all inclusion criteria and do not have exclusion criteria) are given informed consent before enrolling the study and randomized into two groups: erector spinae plane block and spinal. Non-invasive blood pressure monitor, electrocardiogram (ECG), and pulse-oxymetry will be set on the subjects in the operation room. Peripheral venous blood samples will be taken for IL-6 examination. All patients will be sedated using Target Controlled Infusion with propofol (Schnider model, effect site) to obtain mild-moderate sedation prior to the block. On Erector Spinae Plane group, single-shot ultrasound guided block will be performed on the operated side with stimuplex 100 mm needle and 25 ml of isobaric bupivacaine 0.5% with epinephrine 1:200.000 will be administered at level Th 9. On the Spinal group, spinal anesthesia will be performed on lateral decubitus position at the level of L3-L4 or L4-L5 and hyperbaric bupivacaine 0.5% 16-18 mg will be given as regimen. Prior to urethral manipulation, all subjects will be given fentanyl iv 50 mcg and sedation with TCI Propofol will be maintained throughout the procedure. Sensory loss was evaluated by performing skin clamping with a scalpel at the level of the incision before the surgery. The ESP block was considered successful in providing surgical anaesthesia when there was no movement and significant changes in vital signs during skin clamping and throughout the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old and above
* ASA 1,2 and 3
* Patient who will undergo elective supine Percutaneous Nephrolithotomy

Exclusion Criteria:

* Patient who does not agree to be included in the study
* BMI <18.5 kg/m2 or > 40 kg/m2
* Patient with single functional kidney
* Patient who is contraindicated for local anesthetics
* Patient who has severe heart disorder
* Patient with communication disability and cognitive disorders
* Patient with chronic pain with history of high opioid consumption and or alcohol addiction
* Pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence conversion to general anesthesia | intraoperatively
  This outcome will be measured based on the concentration of propofol needed throughout the surgery. If the concentration of propofol exceeds 3.5 mcg/ml, anesthesia will be converted to a general anesthesia.

SECONDARY OUTCOMES:
Interleukin -6 plasma concentration | 24 hours after surgery
  Interleukin 6 will be measured 3 times, before surgery, 6 hours after surgery and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Pry P Pryambodho, Doctor, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided